CLINICAL TRIAL: NCT02487498
Title: A Multi-center, Randomized, Double-blind, Double-dummy, Active Controlled, Two-period Cross-over Study to Assess the Efficacy, Safety and Tolerability of Indacaterol Maleate/Glycopyrronium Bromide Compared to Umeclidinium Bromide/Vilanterol in COPD Patients With Moderate to Severe Airflow Limitation.
Brief Title: Efficacy and Safety Study of Indacaterol Maleate/Glycopyrronium Bromide in Chronic Obstructive Pulmonary Disease (COPD) Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CQVA149A2350
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol-glycopyrronium combination; GSK573719; vilanterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QVA149 (Experimental): QVA149 capsules for inhalation, delivered via QVA149 SDDPI
  Interventions: Drug: QVA149; Drug: Placebo (umeclidinium/vilanterol )
- Umeclidinium/vilanterol (Experimental): Umeclidinium/vilanterol for inhalation, delivered via ELLIPTA® inhaler
  Interventions: Drug: Umeclidinium/vilanterol; Drug: Placebo (QVA149)

INTERVENTIONS:
Drug: QVA149 — QVA149 capsules for inhalation, delivered via QVA149 SDDPI
  Arms: QVA149
Drug: Umeclidinium/vilanterol — Umeclidinium/vilanterol for inhalation, delivered via ELLIPTA® inhaler
  Arms: Umeclidinium/vilanterol
Drug: Placebo (umeclidinium/vilanterol ) — Matching Placebo to umeclidinium/vilanterol for inhalation, delivered via ELLIPTA® inhaler
  Arms: QVA149
Drug: Placebo (QVA149) — Matching Placebo to QVA149 capsules for inhalation, delivered via QVA149 SDDPI
  Arms: Umeclidinium/vilanterol

SUMMARY:
The purpose of this study is to demonstrate that the efficacy of the combination product QVA149 is similar to the efficacy of the combination product umeclidinium/vilanterol on a pre-specified endpoint of FEV1 AUC0-24h while maintaining an acceptable safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged ≥40 yrs
* Smoking history of at least 10 pack years
* Diagnosis of stable Chronic Obstructive Pulmonary Disease (COPD) as classified by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines, 2015)
* Post-bronchodilator Forced Expiratory Volume in 1 Second (FEV1)< 80% and ≥ 30% of the predicted normal value and post-bronchodilator FEV1/FVC (forced vital capacity) <70%
* Modified Medical Research Council questionnaire grade of 2 or higher

Exclusion Criteria:

* Patients who have had a respiratory tract infection within 4 weeks prior to Visit 1
* Patients with concomitant pulmonary disease
* Patients with a history of asthma
* Any patient with lung cancer or a history of lung cancer
* Patients with a history of certain cardiovascular co-morbid conditions
* Patients with a known history and diagnosis of alpha-1 antitrypsin deficiency
* Patients in the active phase of a supervised pulmonary rehabilitation program
* Patients contraindicated for inhaled anticholinergic agents and β2 agonists
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2015-07-27 (Actual); Primary Completion 2016-09-06 (Actual); Study Completion 2016-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (48):
  - Novartis Investigative Site, Anaheim, California
  - Novartis Investigative Site, Escondido, California
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Chiefland, Florida
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Winter Park, Florida
  - Novartis Investigative Site, Florence, Kentucky
  - Novartis Investigative Site, Owensboro, Kentucky
  - Novartis Investigative Site, North Dartmouth, Massachusetts
  - Novartis Investigative Site, Livonia, Michigan
  - Novartis Investigative Site, Saint Charles, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Skillman, New Jersey
  - Novartis Investigative Site, Gastonia, North Carolina
  - Novartis Investigative Site, Monroe, North Carolina
  - Novartis Investigative Site, New Bern, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Shelby, North Carolina
  - Novartis Investigative Site, Wilmington, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Eugene, Oregon
  - Novartis Investigative Site, Pottstown, Pennsylvania
  - Novartis Investigative Site, Anderson, South Carolina
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Easley, South Carolina
  - Novartis Investigative Site, Fort Mill, South Carolina
  - Novartis Investigative Site, Gaffney, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Mt. Pleasant, South Carolina
  - Novartis Investigative Site, Rock Hill, South Carolina
  - Novartis Investigative Site, Seneca, South Carolina
  - Novartis Investigative Site, Simpsonville, South Carolina
  - Novartis Investigative Site, Spartanburg, South Carolina
  - Novartis Investigative Site, Union, South Carolina
  - Novartis Investigative Site, Amarillo, Texas
  - Novartis Investigative Site, Boerne, Texas
  - Novartis Investigative Site, El Paso, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Kingwood, Texas
  - Novartis Investigative Site, Plano, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Greenfield, Wisconsin

REFERENCES:
- [Derived] Kerwin E, Ferguson GT, Sanjar S, Goodin T, Yadao A, Fogel R, Maitra S, Sen B, Ayers T, Banerji D. Dual Bronchodilation with Indacaterol Maleate/Glycopyrronium Bromide Compared with Umeclidinium Bromide/Vilanterol in Patients with Moderate-to-Severe COPD: Results from Two Randomized, Controlled, Cross-over Studies. Lung. 2017 Dec;195(6):739-747. doi: 10.1007/s00408-017-0055-9. Epub 2017 Oct 9. PMID 28993871

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to 1 of 2 sequences in a 1:1 ratio.
Groups:
- First QVA149, Then Umeclidinium/Vilanterol: Participants received QVA149 27.5/12.5 ug via inhalation twice daily (b.i.d.) for 12 weeks. Then after 3 weeks washout, participants received Umeclidinium/vilanterol 62.5/25 ug via inhalation once daily for 12 weeks.
- First Umeclidinium/Vilanterol, Then QVA149: Participants received Umeclidinium/vilanterol 62.5/25 ug via inhalation once daily for 12 weeks. Then after 3 weeks washout, participants received QVA149 27.5/12.5 ug via inhalation twice daily (b.i.d.) for 12 weeks.
Period: Period: Period 1
Arm/Group | First QVA149, Then Umeclidinium/Vilanterol | First Umeclidinium/Vilanterol, Then QVA149
Started | 178 | 177
Completed | 172 | 166
Not Completed | 6 | 11
Not completed — Adverse Event | 2 | 4
Not completed — Subject/guardian decision | 2 | 4
Not completed — Lost to Follow-up | 0 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Protocol deviation | 1 | 0
Period: Period: Washout
Arm/Group | First QVA149, Then Umeclidinium/Vilanterol | First Umeclidinium/Vilanterol, Then QVA149
Started | 172 | 166
Completed | 170 | 159
Not Completed | 2 | 7
Not completed — Subject/guardian decision | 0 | 5
Not completed — Lack of Efficacy | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Non-compliance with study treatment | 0 | 1
Period: Period: Period 2
Arm/Group | First QVA149, Then Umeclidinium/Vilanterol | First Umeclidinium/Vilanterol, Then QVA149
Started | 170 | 159
Completed | 164 | 154
Not Completed | 6 | 5
Not completed — Adverse Event | 2 | 2
Not completed — Subject/guardian decision | 2 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 0 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Since this is a cross-over design study, all participants were randomized to receive both treatments, either in sequence QVA/UV or sequence UV/QVA. Therefore, the baseline characteristics are reported as overall participants.
Groups:
- Overall Participants: Participants received QVA149 27.5/12.5 ug via inhalation twice daily (b.i.d.) for 12 weeks and Umeclidinium/vilanterol 62.5/25 ug via inhalation once daily for 12 weeks.
Arm/Group | Overall Participants
Number analyzed (Participants) | 355
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (8.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163
  Male | 192

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume (FEV1) Area Under the Curve (AUC) 0-24h
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time over an entire day (AUC 0-24h). A positive change from baseline indicates improvement.
Time Frame: baseline, 0 to 24 hours post-dose at week 12
Population: The full analysis, which included all randomized patients who received at least one dose of double-blind treatment, was considered for the analysis. Only participants with a value at both baseline and the post-baseline time point were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | First QVA149, Then Umeclidinium/Vilanterol | First Umeclidinium/Vilanterol, Then QVA149
Number analyzed (Participants) | 319 | 326
Liters | 0.1846 (0.01193) | 0.2028 (0.01188)
Statistical Analysis 1: Comparison: First QVA149, Then Umeclidinium/Vilanterol vs First Umeclidinium/Vilanterol, Then QVA149; Ho: QVA149 27.5/12.5 μg b.i.d. is inferior to umeclidinium/vilanterol 62.5/25 μg q.d; Ha: QVA149 27.5/12.5 μg b.i.d. is non-inferior to umeclidinium/vilanterol 62.5/25 μg q.d; Test type: Non-Inferiority or Equivalence — Non-inferiority was demonstrated if the lower limit (LL) of the 97.5% one -sided confidence interval (CI) > -20 mL; p = 0.415, Linear Mixed Model; Mean Difference (Net) = -0.0182, 95% CI 2-sided [-0.0342 to -0.0023], Standard Error of Mean 0.00813

2. Secondary Outcome: Change From Baseline in Forced Expiratory Volume (FEV1) Area Under the Curve (AUC) 0-24h
Description: as for outcome 1
Time Frame: baseline, 0 to 24 hours post-dose at week 12
Population: The full analysis, which included all randomized patients who received at least one dose of double-blind treatment, was considered for the analysis. Only participants with a value at both baseline and post-baseline time point were included in the analysis
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | First QVA149, Then Umeclidinium/Vilanterol | First Umeclidinium/Vilanterol, Then QVA149
Number analyzed (Participants) | 319 | 326
Liters | 0.1846 (0.01193) | 0.2028 (0.01188)
Statistical Analysis 1: Comparison: First QVA149, Then Umeclidinium/Vilanterol vs First Umeclidinium/Vilanterol, Then QVA149; Test type: Superiority or Other; Mean Difference (Net) = -0.0182, 95% CI 2-sided [-0.0342 to -0.0023], Standard Error of Mean 0.00813

3. Secondary Outcome: Superiority of QVA149 Compared to Umeclidinium/Vilanterol in Terms of Change From Baseline in Trough FEV1 (Mean of 23h 15 Minutes and 23 h 45 Minutes Post Previous Morning Dose)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 15 minutes and 23 hours 45 minutes post-dose for each treatment.
Time Frame: baseline, 23 hours 15 minutes and 23 hours 45 minutes post previous morning dose at week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | First QVA149, Then Umeclidinium/Vilanterol | First Umeclidinium/Vilanterol, Then QVA149
Number analyzed (Participants) | 312 | 312
Liters | 0.1676 (0.01112) | 0.1767 (0.01111)
Statistical Analysis 1: Comparison: First QVA149, Then Umeclidinium/Vilanterol vs First Umeclidinium/Vilanterol, Then QVA149; Test type: Superiority or Other; Mean Difference (Net) = -0.0091, 95% CI 2-sided [-0.0313 to 0.0131], Standard Error of Mean 0.01132

4. Secondary Outcome: Change From Baseline in FEV1 AUC 12-24h
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time over 12 hours (AUC 12-24h).
Time Frame: baseline, 12 hours to 24 hours post-dose at week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | First QVA149, Then Umeclidinium/Vilanterol | First Umeclidinium/Vilanterol, Then QVA149
Number analyzed (Participants) | 317 | 323
Liters | 0.1625 (0.01216) | 0.1539 (0.01210)
Statistical Analysis 1: Comparison: First QVA149, Then Umeclidinium/Vilanterol vs First Umeclidinium/Vilanterol, Then QVA149; Test type: Superiority or Other; Mean Difference (Net) = 0.0086, 95% CI 2-sided [-0.0086 to 0.0258], Standard Error of Mean 0.00874

5. Secondary Outcome: Change From Baseline in FEV1 AUC 0-12h
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time over 12 hours (AUC 0-12h).
Time Frame: baseline, 0 to 12 hours post-dose at week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | First QVA149, Then Umeclidinium/Vilanterol | First Umeclidinium/Vilanterol, Then QVA149
Number analyzed (Participants) | 319 | 326
Liters | 0.2077 (0.01082) | 0.2496 (0.01075)

6. Secondary Outcome: Change From Baseline in FEV1 AUC 0-4h, AUC 4-8h, AUC 8-12h, AUC 12-16h, AUC 16-20h and AUC 20-24h
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time over 4 hour intervals FEV1 AUC 0-4h, AUC 4-8h, AUC 8-12h, AUC 12-16h, AUC 16-20h and AUC 20-24h.
Time Frame: baseline, 12 weeks
Population: The full analysis, which included all randomized patients who received at least one dose of double-blind treatment, was considered for the analysis. Only participants with a value at both baseline and the post-baseline time points were included in the analysis
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | First QVA149, Then Umeclidinium/Vilanterol | First Umeclidinium/Vilanterol, Then QVA149
Number analyzed (Participants) | 337 | 347
Liter
  0-4h: number analyzed (Participants) | 318 | 322
  0-4h | 0.2663 (0.01082) | 0.2938 (0.01077)
  4-8h: number analyzed (Participants) | 316 | 325
  4-8h | 0.1970 (0.01132) | 0.2519 (0.01123)
  8-12h: number analyzed (Participants) | 312 | 322
  8-12h | 0.1513 (0.01143) | 0.2015 (0.01132)
  12-16h: number analyzed (Participants) | 313 | 320
  12-16h | 0.2120 (0.01292) | 0.1842 (0.01285)
  16-20h: number analyzed (Participants) | 314 | 318
  16-20h | 0.1383 (0.01292) | 0.1340 (0.01287)
  20-24h: number analyzed (Participants) | 313 | 319
  20-24h | 0.1374 (0.01197) | 0.1445 (0.01190)

7. Secondary Outcome: QVA149 Compared to Umeclidinium/Vilanterol in Terms of Change From Baseline in Pre-dose Trough FEV1 (Mean of 15 Minutes and 45 Minutes Pre Morning Dose)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Pre-dose trough FEV1 was defined as the average of measurements made 15 minutes and 45 minutes pre morning dose for each treatment.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | First QVA149, Then Umeclidinium/Vilanterol | First Umeclidinium/Vilanterol, Then QVA149
Number analyzed (Participants) | 319 | 326
Liters | 0.1827 (0.01183) | 0.2043 (0.01177)

8. Secondary Outcome: QVA149 Compared to Umeclidinium/Vilanterol in Terms of Change From Baseline in FEV1 at Any Time Point
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards.
Time Frame: Day 1 (5min, 15min, 30min, hours 1, 2, 4, 8, 11h 55min, 23h 15min, 23h 45min); week 6 (-45min, -15min); week 12 (-45min, -15min, 5min, 15min, 30min, hours 1, 2, 4, 8, 11h 55min, 12h 5min, 12h 15min, 12h 30min, 13, 14, 16, 20, 23h 15min, 23h 45min)
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | First QVA149, Then Umeclidinium/Vilanterol | First Umeclidinium/Vilanterol, Then QVA149
Number analyzed (Participants) | 337 | 347
Liters
  Day 1, 5 minutes: number analyzed (Participants) | 323 | 332
  Day 1, 5 minutes | 0.1134 (0.00996) | 0.1117 (0.00984)
  Day 1, 15 minutes: number analyzed (Participants) | 308 | 332
  Day 1, 15 minutes | 0.1448 (0.01081) | 0.1591 (0.01053)
  Day 1, 30 minutes: number analyzed (Participants) | 327 | 335
  Day 1, 30 minutes | 0.1630 (0.01080) | 0.1836 (0.01071)
  Day 1, 1 hour: number analyzed (Participants) | 326 | 336
  Day 1, 1 hour | 0.1742 (0.01133) | 0.2000 (0.01121)
  Day 1, 2 hours: number analyzed (Participants) | 322 | 336
  Day 1, 2 hours | 0.1723 (0.01152) | 0.2138 (0.01136)
  Day 1, 4 hours: number analyzed (Participants) | 323 | 335
  Day 1, 4 hours | 0.1487 (0.01179) | 0.2168 (0.01165)
  Day 1, 8 hours: number analyzed (Participants) | 320 | 332
  Day 1, 8 hours | 0.0908 (0.01160) | 0.1781 (0.01145)
  Day 1, 11 hours 55 minutes: number analyzed (Participants) | 307 | 320
  Day 1, 11 hours 55 minutes | 0.0521 (0.01203) | 0.1537 (0.01185)
  Day 1, 23 hours 15 minutes: number analyzed (Participants) | 313 | 319
  Day 1, 23 hours 15 minutes | 0.1422 (0.01109) | 0.1573 (0.01099)
  Day 1, 23 hours 45 minutes: number analyzed (Participants) | 317 | 325
  Day 1, 23 hours 45 minutes | 0.1702 (0.01156) | 0.1821 (0.01145)
  Week 6, -45 minutes: number analyzed (Participants) | 314 | 323
  Week 6, -45 minutes | 0.1819 (0.01197) | 0.2071 (0.01188)
  Week 6, -15 minutes: number analyzed (Participants) | 307 | 320
  Week 6, -15 minutes | 0.2111 (0.01225) | 0.2343 (0.01214)
  Week 12, -45 minutes: number analyzed (Participants) | 316 | 321
  Week 12, -45 minutes | 0.1750 (0.01195) | 0.1957 (0.01191)
  Week 12, -15 minutes: number analyzed (Participants) | 317 | 321
  Week 12, -15 minutes | 0.1914 (0.01217) | 0.2112 (0.01214)
  Week 12, 5 minutes: number analyzed (Participants) | 303 | 307
  Week 12, 5 minutes | 0.2421 (0.01020) | 0.2563 (0.01015)
  Week 12, 15 minutes: number analyzed (Participants) | 305 | 306
  Week 12, 15 minutes | 0.2681 (0.01086) | 0.2865 (0.01084)
  Week 12, 30 minutes: number analyzed (Participants) | 313 | 318
  Week 12, 30 minutes | 0.2819 (0.01097) | 0.2940 (0.01090)
  Week 12, 1 hour: number analyzed (Participants) | 313 | 319
  Week 12, 1 hour | 0.2919 (0.01149) | 0.3053 (0.01141)
  Week 12, 2 hours: number analyzed (Participants) | 309 | 317
  Week 12, 2 hours | 0.2740 (0.01168) | 0.2994 (0.01158)
  Week 12, 4 hours: number analyzed (Participants) | 312 | 317
  Week 12, 4 hours | 0.2316 (0.01192) | 0.2823 (0.01185)
  Week 12, 8 hours: number analyzed (Participants) | 306 | 313
  Week 12, 8 hours | 0.1631 (0.01176) | 0.2201 (0.01167)
  Week 12, 11 hours 55 minutes: number analyzed (Participants) | 281 | 315
  Week 12, 11 hours 55 minutes | 0.1320 (0.01236) | 0.1812 (0.01193)
  Week 12, 12 hours 5 minutes: number analyzed (Participants) | 304 | 312
  Week 12, 12 hours 5 minutes | 0.1974 (0.01375) | 0.1893 (0.01364)
  Week 12, 12 hours 15 minutes: number analyzed (Participants) | 300 | 306
  Week 12, 12 hours 15 minutes | 0.2107 (0.01375) | 0.1959 (0.01368)
  Week 12, 12 hours 30 minutes: number analyzed (Participants) | 303 | 307
  Week 12, 12 hours 30 minutes | 0.2296 (0.01355) | 0.1934 (0.01350)
  Week 12, 13 hours: number analyzed (Participants) | 299 | 310
  Week 12, 13 hours | 0.2341 (0.01376) | 0.1953 (0.01364)
  Week 12, 14 hours: number analyzed (Participants) | 296 | 310
  Week 12, 14 hours | 0.2308 (0.01372) | 0.1966 (0.01357)
  Week 12, 16 hours: number analyzed (Participants) | 303 | 304
  Week 12, 16 hours | 0.1705 (0.01382) | 0.1582 (0.01381)
  Week 12, 20 hours: number analyzed (Participants) | 309 | 308
  Week 12, 20 hours | 0.1078 (0.01338) | 0.1158 (0.01338)
  Week 12, 23 hours 15 minutes: number analyzed (Participants) | 307 | 308
  Week 12, 23 hours 15 minutes | 0.1573 (0.01117) | 0.1648 (0.01115)
  Week 12, 23 hours 45 minutes: number analyzed (Participants) | 312 | 308
  Week 12, 23 hours 45 minutes | 0.1798 (0.01163) | 0.1892 (0.01167)

9. Secondary Outcome: QVA149 Compared to Umeclidinium/Vilanterol in Terms of Change From Baseline in Forced Vital Capacity (FVC) at Any Time Point
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards.
Time Frame: Day 1 (5min, 15min, 30 min, hours 1, 2, 4, 8, 11h 55min, 23h 15min, 23h 45min); week 6 (-45min, -15min); week 12 (-45min, -15min, 5min, 15min, 30min, hours 1, 2, 4, 8, 11h 55min, 12h 5min, 12h 15min, 12h 30min, 13, 14, 16, 20, 23h 15min, 23h 45min)
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | First QVA149, Then Umeclidinium/Vilanterol | First Umeclidinium/Vilanterol, Then QVA149
Number analyzed (Participants) | 337 | 347
Liters
  Day 1, 5 minutes: number analyzed (Participants) | 323 | 332
  Day 1, 5 minutes | 0.1994 (0.01672) | 0.2054 (0.01655)
  Day 1, 15 minutes: number analyzed (Participants) | 308 | 332
  Day 1, 15 minutes | 0.2454 (0.01764) | 0.2589 (0.01724)
  Day 1, 30 minutes: number analyzed (Participants) | 327 | 335
  Day 1, 30 minutes | 0.2734 (0.01806) | 0.3028 (0.01792)
  Day 1, 1 hour: number analyzed (Participants) | 326 | 336
  Day 1, 1 hour | 0.2841 (0.01937) | 0.3136 (0.01917)
  Day 1, 2 hours: number analyzed (Participants) | 322 | 336
  Day 1, 2 hours | 0.2708 (0.01928) | 0.3334 (0.01904)
  Day 1, 4 hours: number analyzed (Participants) | 323 | 335
  Day 1, 4 hours | 0.2333 (0.01914) | 0.3405 (0.01892)
  Day 1, 8 hours: number analyzed (Participants) | 320 | 332
  Day 1, 8 hours | 0.1728 (0.01923) | 0.3067 (0.01900)
  Day 1, 11 hours 55 minutes: number analyzed (Participants) | 307 | 320
  Day 1, 11 hours 55 minutes | 0.1291 (0.01971) | 0.2654 (0.01944)
  Day 1, 23 hours 15 minutes: number analyzed (Participants) | 313 | 319
  Day 1, 23 hours 15 minutes | 0.2387 (0.01789) | 0.2363 (0.01775)
  Day 1, 23 hours 45 minutes: number analyzed (Participants) | 317 | 325
  Day 1, 23 hours 45 minutes | 0.2821 (0.01886) | 0.2940 (0.01868)
  Week 6, -45 minutes: number analyzed (Participants) | 314 | 323
  Week 6, -45 minutes | 0.2666 (0.01958) | 0.3045 (0.01942)
  Week 6, -15 minutes: number analyzed (Participants) | 307 | 320
  Week 6, -15 minutes | 0.2860 (0.01963) | 0.3372 (0.01943)
  Week 12, -45 minutes: number analyzed (Participants) | 316 | 321
  Week 12, -45 minutes | 0.2264 (0.01956) | 0.2737 (0.01947)
  Week 12, -15 minutes: number analyzed (Participants) | 317 | 321
  Week 12, -15 minutes | 0.2468 (0.01949) | 0.2844 (0.01943)
  Week 12, 5 minutes: number analyzed (Participants) | 303 | 307
  Week 12, 5 minutes | 0.3386 (0.01711) | 0.3489 (0.01701)
  Week 12, 15 minutes: number analyzed (Participants) | 305 | 306
  Week 12, 15 minutes | 0.3616 (0.01771) | 0.3811 (0.01768)
  Week 12, 30 minutes: number analyzed (Participants) | 313 | 318
  Week 12, 30 minutes | 0.3796 (0.01830) | 0.4019 (0.01821)
  Week 12, 1 hour: number analyzed (Participants) | 313 | 319
  Week 12, 1 hour | 0.3935 (0.01962) | 0.4085 (0.01949)
  Week 12, 2 hours: number analyzed (Participants) | 309 | 317
  Week 12, 2 hours | 0.3708 (0.01953) | 0.4050 (0.01937)
  Week 12, 4 hours: number analyzed (Participants) | 312 | 317
  Week 12, 4 hours | 0.3261 (0.01933) | 0.3845 (0.01924)
  Week 12, 8 hours: number analyzed (Participants) | 306 | 313
  Week 12, 8 hours | 0.2259 (0.01950) | 0.3152 (0.01936)
  Week 12, 11 hours 55 minutes: number analyzed (Participants) | 281 | 315
  Week 12, 11 hours 55 minutes | 0.1900 (0.02023) | 0.2749 (0.01956)
  Week 12, 12 hours 5 minutes: number analyzed (Participants) | 304 | 312
  Week 12, 12 hours 5 minutes | 0.2817 (0.02157) | 0.2711 (0.02141)
  Week 12, 12 hours 15 minutes: number analyzed (Participants) | 300 | 306
  Week 12, 12 hours 15 minutes | 0.3010 (0.02177) | 0.2762 (0.02165)
  Week 12, 12 hours 30 minutes: number analyzed (Participants) | 303 | 307
  Week 12, 12 hours 30 minutes | 0.3279 (0.02155) | 0.2786 (0.02146)
  Week 12, 13 hours: number analyzed (Participants) | 299 | 310
  Week 12, 13 hours | 0.3381 (0.02210) | 0.2909 (0.02189)
  Week 12, 14 hours: number analyzed (Participants) | 296 | 310
  Week 12, 14 hours | 0.3445 (0.02233) | 0.2984 (0.02208)
  Week 12, 16 hours | 0.2496 (0.02191) | 0.2514 (0.02188)
  Week 12, 20 hours: number analyzed (Participants) | 309 | 308
  Week 12, 20 hours | 0.1600 (0.02168) | 0.1845 (0.02169)
  Week 12, 23 hours 15 minutes: number analyzed (Participants) | 307 | 308
  Week 12, 23 hours 15 minutes | 0.2026 (0.01802) | 0.2251 (0.01800)
  Week 12, 23 hours 45 minutes: number analyzed (Participants) | 312 | 308
  Week 12, 23 hours 45 minutes | 0.2415 (0.01897) | 0.2662 (0.01903)

ADVERSE EVENTS:
Description: Since this is a cross-over design study, all patients were randomized to receive both treatments, either in sequence QVA/UV or sequence UV/QVA. The number of patients on each treatment does not add up to the total number of patients.
Groups:
- QVA 27.5/12.5 Bid: QVA149 capsules for inhalation, delivered via QVA149 SDDPI
- U/V 62.5/25 od: Umeclidinium/vilanterol for inhalation, delivered via ELLIPTA® inhaler
- All Patients: All Patients
Arm/Group | QVA 27.5/12.5 Bid | U/V 62.5/25 od | All Patients
Serious Adverse Events (participants affected / at risk) | 17/337 | 10/347 | 26/355
Other Adverse Events (participants affected / at risk) | 78/337 | 89/347 | 140/355
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA 27.5/12.5 Bid (N=337) | U/V 62.5/25 od (N=347) | All Patients (N=355)
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 2 | 0 | 2
Myocardial infarction (Cardiac disorders) | 1 | 1 | 2
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 2 | 3
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cervix carcinoma stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 10
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 1 | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0 | 1
Vascular insufficiency (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVA 27.5/12.5 Bid (N=337) | U/V 62.5/25 od (N=347) | All Patients (N=355)
Acute sinusitis (Infections and infestations) | 3 | 1 | 4
Bronchitis (Infections and infestations) | 11 | 6 | 16
Gastroenteritis viral (Infections and infestations) | 3 | 1 | 4
Lower respiratory tract infection (Infections and infestations) | 4 | 3 | 7
Nasopharyngitis (Infections and infestations) | 3 | 4 | 7
Oral candidiasis (Infections and infestations) | 4 | 2 | 6
Sinusitis (Infections and infestations) | 6 | 5 | 11
Upper respiratory tract infection (Infections and infestations) | 5 | 8 | 13
Upper respiratory tract infection bacterial (Infections and infestations) | 4 | 7 | 9
Viral upper respiratory tract infection (Infections and infestations) | 3 | 8 | 11
Laceration (Injury, poisoning and procedural complications) | 2 | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5
Headache (Nervous system disorders) | 2 | 3 | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 50 | 51 | 89
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety